CLINICAL TRIAL: NCT03968302
Title: ADDITION OF BISMUTH TO THE STANDARD TRIPLE THERAPY FOR HELICOBACTER PYLORI ERADICATION: A RANDOMIZED CONTROLLED STUDY
Brief Title: ADDITION OF BISMUTH TO THE STANDARD TRIPLE THERAPY FOR HELICOBACTER PYLORI ERADICATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Muhammad Asim, GI FELLOW, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZiauddinU
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: H pylori; eradication; amoxicillin; clarithromycin; esomeprazole; colloidal bismuth subcitrate

STUDY DESIGN:
Intervention Model Description: PARALLEL ASSIGNMENT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A (Experimental): The triple regimen, amoxicillin 1 gm twice a day, clarithromycin 500 mg twice a day and omeprazole 40 mg twice a day
  Interventions: Drug: ARM A Triple therapy for helicobacter pylori
- ARM B (Experimental): The quadruple regimen,amoxicillin 1 gm twice a day, clarithromycin 500 mg twice a day, omeprazole 40 mg twice a day dose and colloidal bismuth subcitrate 240 mg twice daily
  Interventions: Drug: ARM B Quadruple therapy for helicobacter pylori

INTERVENTIONS:
Drug: ARM A Triple therapy for helicobacter pylori — The triple regimen was defined as a combination of amoxicillin 1 gm twice a day, clarithromycin 500 mg twice a day and omeprazole is given in 40 mg twice a day dose.
  Arms: ARM A
Drug: ARM B Quadruple therapy for helicobacter pylori — Quadruple therapy included colloidal bismuth subcitrate 240 mg twice daily,amoxicillin 1 gm twice a day, clarithromycin 500 mg twice a day and omeprazole is given in 40 mg twice a day dose.
  Arms: ARM B

SUMMARY:
H pylori is an important cause of chronic gastritis and other complications. There is a decline in eradication rate for H pylori owing to multiple factors including drug resistance. We compare the effect of the addition of bismuth to the standard triple therapy in a randomized control trial.

Subjects were randomized into two arms. Arm A received triple therapy including amoxicillin, clarithromycin, and omeprazole and Arm B received quadruple therapy adding colloidal bismuth subcitrate. Both arms received treatment for two weeks.

DETAILED DESCRIPTION:
The study is a 2-arm, prospective, randomized, non-inferiority, unblinded, parallel design trial. The primary end point is post-treatment result after triple or quadruple therapy. Secondary endpoints included the nature and frequency of side effects compared between the two arms. The study protocol was approved by the ethical review committee of the university.

Patients with dyspeptic symptoms who had H pylori infection, diagnosed through positive Stool for H pylori antigen or presence of H. pylori organism in the histopathology of gastric mucosal biopsy, attending outpatient department of two campuses of the University Hospital were included in this study.. Group A received standard triple therapy for H. pylori eradication for a total 14 days and group B received bismuth-based quadruple therapy for H pylori eradication for the same period. The triple regimen was defined as a combination of amoxicillin 1 gm twice a day, clarithromycin 500 mg twice a day and omeprazole is given in 40 mg twice a day dose. Quadruple therapy included colloidal bismuth subcitrate 240 mg twice daily, in addition. H. Pylori status was checked routinely after 6 weeks by Stool sampling for H, pylori antigen. Subjects were counseled to stop taking PPI or any antibiotic 2 weeks before stool H. pylori antigen testing. Eradication of H pylori was defined as lack of detection of H pylori antigen in the stool via ELISA method after triple or quadruple therapy.

ELIGIBILITY:
Inclusion Criteria:

Patients with dyspeptic symptoms who had H pylori infection, diagnosed through positive Stool for H pylori antigen or presence of H. pylori organism in the histopathology of gastric mucosal biopsy, attending outpatient department of two campuses of the University Hospital were included in this study

Exclusion Criteria:

Exclusion criteria were patients with age less than 12 years, age more than 80 years, recent antibiotic use, and treatment-experienced patients, where H. pylori couldn't eradicate after treatment, chronic illnesses with multiple comorbid for example, chronic liver disease, chronic kidney disease or terminal illness etc, pregnancy and allergy to any of the regimen components.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
POST H PYLORI TREATMENT RESULTS | 2 months
  The primary end point was post-treatment result after triple or quadruple therapy

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD ASIM, MBBS, Principal Investigator — ZIAUDDIN UNIVERSITY HOSPITAL; KHURRAM BAQAI, FCPS, Principal Investigator — Ziauddin University; ZAIGHAM ABBAS, FCPS, Study Chair — Ziauddin University
Locations (1):
- Ziauddin University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No